CLINICAL TRIAL: NCT06192186
Title: The Safety and Efficacy of Adebrelimab Combined With SOX Regimen in Preoperative Neoadjuvant Therapy for Locally Advanced Gastric Adenocarcinoma Patients (ASOG-01)
Brief Title: Adebrelimab Combined With SOX Regimen in Preoperative Neoadjuvant Transformation Therapy for Locally Advanced Gastric Adenocarcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yang Jianjun, PhD (Other)
Responsible Party: Sponsor-Investigator, Yang Jianjun, PhD, Professor from Xijing Hospital, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASOG-01
Record Dates: First submitted 2023-11-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Locally Advanced Gastric Adenocarcinoma
Keywords: Adebrelimab; SOX regimen; Preoperative neoadjuvant transformation therapy; Locally advanced gastric adenocarcinoma; Randomized controlled clinical trial
MeSH Terms: interventions — Clinical Protocols

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This study is a double-blind design, which blinds both the researcher and the patient. Considering that adebrelimab is administered by injection and the solvent is a 5% glucose solution, therefore, the control group will use 5% glucose solution as placebo. They are not easily distinguishable in appearance, so patients can be blinded. During the research process, patient grouping information will be randomly extracted by Jialin Luo, and kept confidential to other researchers (other members who responsible for follow-up and analysis) until unblinding. Meanwhile, Jialin Luo did not participate in the follow-up and statistical analysis of patients after medication.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adebrelimab combined with SOX regimen (Experimental): Adebrelimab combined with SOX regimen preoperatively used 3 cycles(stop adebrelimab and S-1/oxaliplatin after 3 cycles and evaluate tumor staging)→ radical surgery (D2) →Postoperative selection of continued medication or cessation of treatment will base on the patient's pathological reports. Surgery should be performed within 3-6 weeks after 3 cycles of preoperative neoadjuvant therapy.
  Interventions: Drug: Adebrelimab combined with SOX regimen
- Placebo combined with SOX (S-1/oxaliplatin) regimen (Active Comparator): Placebo combined with SOX (S-1/oxaliplatin) regimen preoperatively used 3 cycles(stop placebo and S-1/oxaliplatin after 3 cycles and evaluate tumor staging)→ radical surgery (D2) →Postoperative selection of continued medication or cessation of treatment will base on the patient's pathological reports. Surgery should be performed within 3-6 weeks after 3 cycles of preoperative neoadjuvant therapy.
  Interventions: Drug: Placebo combined with SOX (S-1/oxaliplatin) regimen

INTERVENTIONS:
Drug: Adebrelimab combined with SOX regimen — Adebrelimab combined with SOX regimen preoperatively used 3 cycles(stop adebrelimab and S-1/oxaliplatin after 3 cycles and evaluate tumor staging)→ radical surgery (D2) →Postoperative selection of continued medication or cessation of treatment will base on the patient's pathological reports. Surgery should be performed within 3-6 weeks after 3 cycles of preoperative neoadjuvant therapy.
  Arms: Adebrelimab combined with SOX regimen
Drug: Placebo combined with SOX (S-1/oxaliplatin) regimen — Placebo combined with SOX (S-1/oxaliplatin) regimen preoperatively used 3 cycles (stop placebo and S-1/oxaliplatin after 3 cycles and evaluate tumor staging) → radical surgery (D2) →Postoperative selection of continued medication or cessation of treatment will base on the patient's pathological reports. Surgery should be performed within 3-6 weeks after 3 cycles of preoperative neoadjuvant therapy.
  Arms: Placebo combined with SOX (S-1/oxaliplatin) regimen

SUMMARY:
Abstract Objective: Adebrelimab is a PD-L1 inhibitor. The aim of this trial is to evaluate the safety and efficacy of adebrelimab combined with SOX regimen for preoperative neoadjuvant therapy in locally advanced gastric adenocarcinoma.

Methods and analysis: This study is a prospective single-center, two-arm, double-blind and randomized controlled clinical trial designed to include 110 patients with locally advanced gastric adenocarcinoma who will be randomly assigned into two groups: experimental group (adebrelimab combined with SOX regimen) (n=55) and control group (SOX regimen) (n=55). The main efficacy indicators are pathological complete response rate (pCR). The secondary efficacy indicators are R0 resection rate, safety indicators (including surgical and drug treatment safety indicators). disease-free survival (DFS) and overall survival (OS).

Ethics: Ethics approval has been obtained from the Ethics Committee at the First Affiliated Hospital (Xijing Hospital) of Air force Military Medical University (KY20232357-F-1).

ELIGIBILITY:
The inclusion criteria is as follows:

Patients are able to and willing to provide written informed consent to participate in the study.

Patients are aged 18-75 years old with an Eastern Cooperative Oncology Group (ECOG) score: 0-1 points and expected survival time ≥ 12 weeks.

Patients are diagnosed with gastric adenocarcinoma by pathological examination and the clinical stage should be clinical stage III (T3-4a/N+M0, T3-4a/N-M0), the tumor of the patients with adenocarcinoma of the gastroesophageal junction should be not involve the dentate line.

Functions of the major organs and bone marrow meet the following criteria within 7 days before treatment: hemoglobin ≥ 90g/L, absolute neutrophil count ≥ 1.5 × 109/L, platelet (PLT) ≥ 80× 109/L, without blood transfusion within 14 days, total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN), Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5x ULN, serum creatinine ≤ 1.5x ULN or creatinine clearance ≥ 60mL/min.

Doppler ultrasound: Left ventricular ejection fraction (LVEF) ≥ lower limit of normal value (50%).

Have not received anti-tumor treatment (such as surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy).

The exclusion criteria is as follows:

Other malignant tumors that have occurred or are currently present within 5 years, excluding cured cervical cancer in situ, non-melanoma skin cancer, and superficial bladder tumors.

Patients who require systemic treatment with corticosteroids (>10mg prednisone equivalent dose per day) or other immunosuppressive drugs within 14 days before the start of treatment.

Patients with significant malnutrition. Patients receiving live/attenuated vaccines during treatment. Patients with any severe and/or uncontrollable diseases, including hypertension who cannot be well controlled with antihypertensive medication (systolic blood pressure ≥ 150mm Hg, diastolic blood pressure ≥ 100mm Hg); grade I or above myocardial ischemia or infarction, arrhythmia (including QTc ≥ 480ms) and ≥ grade 2 congestive heart failure (New York Heart Association (NYHA) classification); severe or uncontrolled active infections (≥ CTCAE2 level infection); renal failure requires hemodialysis or peritoneal dialysis; patients with a history of immune deficiency, including those who are HIV positive or suffer from other acquired or congenital immune deficiency diseases; poor blood glucose control in diabetes patients (fasting blood glucose (FBG)>10mmol/L); patients with epileptic seizures who require treatment; patients with previous and current history of interstitial lung disease, pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe impairment of lung function, etc., may interfere with the detection and management of suspected drug-related pulmonary toxicity; patients with gastrointestinal bleeding, perforation, or obstruction.

Patients with any bleeding event ≥ CTCAE3 level within the first 4 weeks of enrollment, as well as patients with unhealed wounds, ulcers, or fractures.

Patients who have experienced arterial/venous thrombosis events within 3 months, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis and pulmonary embolism.

Patients who are preparing to undergo or have previously received allogeneic organ or bone marrow transplantation.

According to the judgment of the researchers, patients with other accompanying diseases that seriously endanger patient safety or affect the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR | 48 months
  pathological complete response rate (pCR)

SECONDARY OUTCOMES:
R0 resection rate | 48 months
  R0 resection rate
AE | 48 months
  the incidence of adverse events (AE)
DFS | 48 months
  disease-free survival
OS | 48 months
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of the Air Force Medical University, Xi'an, China

IPD SHARING:
Plan to Share IPD: No